CLINICAL TRIAL: NCT01138150
Title: Ictal and Interictal Inflammatory Markers in Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Toledo Health Science Campus (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: GSK112035; NCT00868322 (obsolete NCT alias)
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Migraine
Keywords: migraine, headache, sumatriptan, naproxen sodium
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — sumatriptan-naproxen; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treximet (Active Comparator): Fourteen participants randomized to receive Treximet (sumatriptan & naproxen) during an acute migraine attack. Blood drawn for immune & inflammatory markers (adipocytokines,cytokines, sex hormones) at different time points - on presentation with moderate to severe migraine pain; then 30 minutes, 1 hour and 2 hours after administration of study drug (Treximet).
  Participants will be offered a traditional headache rescue medicine at 2 hours after administration of Treximet if participant still reports moderate to severe pain and desires further treatment. Rescue medicine may include the following: prochlorperazine 10 mg IV preceded by diphenhydramine 25 mg IV/PO or metoclopramide 10 mg IV preceded by diphenhydramine 25 mg IV/PO or Toradol 30 mg IV to be determined by the physician.
  Interventions: Drug: Treximet
- Sugar Pill (Placebo Comparator): Fourteen participants randomized to receive placebo during an acute migraine attack. Blood is drawn for immune & inflammatory markers (adipocytokines,cytokines), sex hormones at different time points - on presentation with moderate to severe migraine pain, then 30 minutes, 1 hour and 2 hours after administration of placebo.
  Participants will be offered a traditional headache rescue medicine at 2 hours after administration of placebo if participant still reports moderate to severe pain and desires further treatment. Rescue medicine may include the following: prochlorperazine 10 mg IV preceded by diphenhydramine 25 mg IV/PO or metoclopramide 10 mg IV preceded by diphenhydramine 25 mg IV/PO or Toradol 30 mg IV to be determined by the physician.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Treximet — One tablet of sumatriptan 85 mg and naproxen sodium 500 mg will be given upon subject presentation with an acute migraine attack and after blood levels have been drawn.
  Other Names: The brand name of sumatriptan/naproxen sodium is Treximet.
  Arms: Treximet
Drug: Placebo — One tablet of a sugar pill will be given upon subject presentation with an acute migraine attack and after blood levels have been drawn.
  Other Names: Sugar Pill
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to evaluate blood levels of several proteins that may be altered in the inflammation associated with migraine headaches. These blood levels will be evaluated in individuals during an acute migraine attack and compared to their levels when pain free. The investigators study hypothesis is that the pro inflammatory proteins in the blood will be greater than the levels of these proteins when evaluated during a pain free period.

DETAILED DESCRIPTION:
Migraine is a common, chronic disorder, which presents with recurrent episodes of disabling headache and affects approximately 12% of American adults.1,2 No biomarkers exist to identify episodic or chronic migraine sufferers; and the diagnosis relies solely on clinical criteria. Further the full pathophysiology of migraine has not been fully delineated, although our understanding of migraine pathophysiology has dramatically improved over the past 15 years. Current theories suggest that migraine is a neurovascular disorder, with the pain of migraine a result of the release of inflammatory neuropeptides from nerve endings in the activated trigeminal system (neurogenic inflammation), ultimately resulting in vasodilation, plasma extravasation and mast cell degranulation.3-6 Several inflammatory markers have been implicated in the pathway resulting in the neurogenic inflammation of migraine including calcitonin gene related peptide (CGRP), substance P (SP), neurokinin A, and multiple cytokines such as interleukin (IL) -1, IL-6 and tumor necrosis-α (TNF-α).5,7-10 More recent research supports that the odds of migraine are increased in those who are obese and that several adipose tissue derived cytokines (adipocytokines) may contribute to the neurogenic inflammation of migraine, including leptin and adiponectin. In one small pilot study of 33 participants evaluating chronic and episodic migraineurs as compared to controls, adiponectin (an adipocytokine) was significantly elevated in chronic migraineurs as compared to controls. A second study reported low levels of another adipocytokine, leptin in episodic migraineurs. However, all of these studies have evaluated only 3 to 4 of cytokines at the same time point and 11 none have evaluated adipocytokines during an acute attack. We hypothesize that obesity-related cytokines contribute to the neurogenic inflammation of migraine and have the potential be useful as biomarkers for episodic and chronic migraine as well as new drug targets for the treatment of migraine. To this end we propose to evaluate serum levels of obesity-related cytokines in migraineurs, ictally (during an acute migraine attack), following treatment with sumatriptan/naproxen sodium (Treximet®) and interictally (at baseline) when pain free.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years of age, migraine

Exclusion Criteria:

* Pregnant or breast-feeding women, presence of cardiovascular or cerebrovascular disorders as well as any known inflammatory, infectious, metabolic, thyroid, renal, cardiovascular or gastrointestinal diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Peterlin, DO, Principal Investigator — The Johns Hopkins University
Locations (1):
- The Johns Hopkins Bayview Headache Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment - December 9 2010 through January 22, 2013.
  Types of location - Neurology Headache Clinic, Internal Medicine Clinics, Gynecology clinic; study flyers placed in the medical offices , Johns Hopkins Community Physicians sites, academic institutions and wellness centers.
Groups:
- Active Drug - Sumatriptan/Naproxen: Participants randomized to sumatriptan/naproxen upon presentation of migraine acute attack
- Placebo: Participants randomized to placebo upon presentation with acute migraine attack.
Period: Overall Study
Arm/Group | Active Drug - Sumatriptan/Naproxen | Placebo
Started | 18 | 18
Completed | 17 | 17
Not Completed | 1 | 1
Not completed — blood unable to be processed | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treximet: Participants randomized to active drug Treximet during acute migraine attack.
- Sugar Pill: Participants randomized to placebo (sugar pill) during acute migraine attack.
- Total: Total of all reporting groups
Arm/Group | Treximet | Sugar Pill | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in the Total Serum Adiponectin (T-ADP)
Description: Change in total serum adiponectin after treatment in responders and non responders
Time Frame: 30 minutes after treatment, 60 minutes after treatment, 120 minutes after treatment
Measure: Mean (95% Confidence Interval); unit: ug/mL
Groups:
- Treatment Responders 30 Minutes After Treatment: Treatment responders are defined as those with a reduction of pain from moderate to severe at T0 (before treatment) to none to mild 30 minutes after treatment with Treximet or sugar pill.
- Treatment Non-Responders 30 Minutes After Treatment: Treatment non-responders are defined as those without a reduction of pain from moderate to severe at T0 (before treatment) to none to mild 30 minutes after after treatment with Treximet or sugar pill.
- Treatment Responders 60 Minutes After Treatment: Treatment responders are defined as those with a reduction of pain from moderate to severe at T0 (before treatment) to none to mild 60 minutes after treatment with Treximet or sugar pill.
- Treatment Non-Responders 60 Minutes After Treatment: Treatment non-responders are defined as those without a reduction of pain from moderate to severe at T0 (before treatment) to none to mild 60 minutes after treatment with Treximet or sugar pill.
- Treatment Responders 120 Minutes After Treatment: Treatment responders are defined as those with a reduction of pain from moderate to severe at T0 (before treatment) to none to mild 120 minutes after treatment with Treximet or sugar pill.
- Treatment Non-Responders: Treatment non-responders are defined as those without a reduction of pain from moderate to severe at T0 (before treatment) to none to mild 120 minutes after treatment with Treximet or sugar pill.
Arm/Group | Treatment Responders 30 Minutes After Treatment | Treatment Non-Responders 30 Minutes After Treatment | Treatment Responders 60 Minutes After Treatment | Treatment Non-Responders 60 Minutes After Treatment | Treatment Responders 120 Minutes After Treatment | Treatment Non-Responders
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 17
ug/mL | -0.96 [-1.84 to -0.08] | 0.25 [-1.85 to 2.37] | -0.97 [-1.85 to -0.08] | 0.29 [-1.88 to 2.46] | -0.98 [-1.88 to -0.08] | 0.24 [-1.95 to 2.44]

2. Secondary Outcome: High Molecular Weight (HMW)-Adiponectin (ADP)
Description: serum HMW-ADP levels after treatment in responders and non responders
Time Frame: 30 minutes after treatment, 60 minutes after treatment, 120 minutes after treatment
Measure: Mean (95% Confidence Interval); unit: ug/mL
Groups:
- Treatment Responders 120 Minutes After Treatment; Treatment Responders 30 Minutes After Treatment; Treatment Responders 60 Minutes After Treatment: Treatment responders were defined as those with a reduction of pain from moderate to severe (>=4/10 on the NRS) at T0 to no to mild (<=3/10 on the NRS) at 120 minutes after treatment with either sumatriptan/naproxen or placebo
- Treatment Non Responders 120 Minutes After Treatment; Treatment Non-Responders 30 Minutes After Treatment; Treatment Non-Responders 60 Minutes After Treatment: Participants without reduction in pain at 120 minutes after treatment
Arm/Group | Treatment Responders 120 Minutes After Treatment | Treatment Non Responders 120 Minutes After Treatment | Treatment Responders 30 Minutes After Treatment | Treatment Non-Responders 30 Minutes After Treatment | Treatment Non-Responders 60 Minutes After Treatment | Treatment Responders 60 Minutes After Treatment
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 17
ug/mL | -0.24 [-0.47 to -0.01] | -0.08 [-0.76 to 0.61] | -0.23 [-0.46 to -0.01] | -0.14 [-0.79 to 0.52] | -0.24 [-0.91 to 0.44] | -0.21 [-0.44 to 0.01]

3. Secondary Outcome: Middle Molecular Weight (MMW)-ADP
Description: serum MMW-ADP levels after treatment in responders and non responders
Time Frame: 30 minutes after treatment, 60 minutes after treatment, 120 minutes after treatment
Measure: Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Treatment Responders 120 Minutes After Treatment | Treatment Non Responders 120 Minutes After Treatment | Treatment Responders 30 Minutes After Treatment | Treatment Non-Responders 30 Minutes After Treatment | Treatment Non-Responders 60 Minutes After Treatment | Treatment Responders 60 Minutes After Treatment
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 17
ug/mL | -0.02 [-0.25 to 0.22] | 0.02 [-0.19 to 0.24] | -0.03 [-0.26 to 0.21] | -0.02 [-0.23 to 0.19] | 0.16 [-0.05 to 0.38] | -0.03 [-0.26 to 0.21]

4. Secondary Outcome: Low Molecular Weight (LMW)-ADP
Description: serum LMW-ADP levels after treatment in responders and non responders
Time Frame: 30 minutes after treatment, 60 minutes after treatment, 120 minutes after treatment
Measure: Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Treatment Responders 120 Minutes After Treatment | Treatment Non Responders 120 Minutes After Treatment | Treatment Responders 30 Minutes After Treatment | Treatment Non-Responders 30 Minutes After Treatment | Treatment Non-Responders 60 Minutes After Treatment | Treatment Responders 60 Minutes After Treatment
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 17
ug/mL | 0.32 [0.03 to 0.60] | -0.43 [-0.75 to -0.11] | 0.15 [-0.13 to 0.42] | -0.25 [-0.57 to 0.06] | -0.45 [-0.77 to -0.14] | 0.11 [-0.17 to 0.39]

5. Secondary Outcome: High Molecular Weight (HMW): T-ADP
Description: serum HMW:T-ADP levels after treatment in responders and non responders
Time Frame: 30 minutes, 60 minutes, 120 minutes after treatment
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Treatment Responders 120 Minutes After Treatment | Treatment Non Responders 120 Minutes After Treatment | Treatment Responders 30 Minutes After Treatment | Treatment Non-Responders 30 Minutes After Treatment | Treatment Non-Responders 60 Minutes After Treatment | Treatment Responders 60 Minutes After Treatment
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 17
ratio | -0.04 [-0.07 to -0.01] | 0.01 [-0.03 to 0.06] | -0.02 [-0.06 to 0.01] | 0.01 [-0.04 to 0.05] | 0.01 [-0.05 to 0.05] | -0.02 [-0.05 to 0.02]

6. Secondary Outcome: Low Molecular Weight (LMW):Total (T)-ADP
Description: serum LMW:T-ADP levels after treatment in responders and non responders
Time Frame: 30 minutes after treatment, 60 minutes after treatment, 120 minutes after treatment
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Treatment Responders 120 Minutes After Treatment | Treatment Non Responders 120 Minutes After Treatment | Treatment Responders 30 Minutes After Treatment | Treatment Non-Responders 30 Minutes After Treatment | Treatment Non-Responders 60 Minutes After Treatment | Treatment Responders 60 Minutes After Treatment
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 17
ratio | 0.04 [0.01 to 0.07] | -0.04 [-0.07 to -0.01] | -0.01 [-0.05 to 0.02] | 0.02 [-0.02 to 0.05] | -0.04 [-0.07 to -0.01] | 0.01 [-0.02 to 0.05]

7. Secondary Outcome: Leptin
Description: serum leptin levels after treatment in responders and non responders
Time Frame: 30 minutes after treatment, 60 minutes after treatment, 120 minutes after treatment
Measure: Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Treatment Responders 120 Minutes After Treatment | Treatment Non Responders 120 Minutes After Treatment | Treatment Responders 30 Minutes After Treatment | Treatment Non-Responders 30 Minutes After Treatment | Treatment Non-Responders 60 Minutes After Treatment | Treatment Responders 60 Minutes After Treatment
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 17
ug/mL | 0.71 [-1.55 to 2.97] | 0.89 [-0.93 to 2.71] | 0.28 [-1.93 to 2.50] | 0.84 [-0.91 to 2.59] | 1.00 [-0.80 to 2.80] | 0.02 [-2.21 to 2.24]

8. Secondary Outcome: Resistin
Description: serum resistin levels after treatment in responders and non responders
Time Frame: 30 minutes after treatment, 60 minutes after treatment, 120 minutes after treatment
Measure: Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Treatment Responders 120 Minutes After Treatment | Treatment Non Responders 120 Minutes After Treatment | Treatment Responders 30 Minutes After Treatment | Treatment Non-Responders 30 Minutes After Treatment | Treatment Non-Responders 60 Minutes After Treatment | Treatment Responders 60 Minutes After Treatment
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 17
ug/mL | -0.95 [-1.83 to -0.07] | -0.97 [-3.95 to 2.00] | -1 [-1.86 to -0.14] | -0.88 [-3.75 to 1.98] | -1.36 [-4.30 to 1.59] | -0.79 [-1.65 to 0.08]

ADVERSE EVENTS:
Groups:
- Treximet: sumatriptan/naproxen sodium: One tablet of sumatriptan 85 mg and naproxen sodium 500 mg will be given upon subject presentation with an acute migraine attack and after blood levels have been drawn.
Arm/Group | Treximet | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No